CLINICAL TRIAL: NCT07028762
Title: Motor Coordination During Catching of a Moving Object in Preschool Children as the Indicator of Motor Development
Brief Title: Evaluation of Catching Skills in Preschoolers With Motor Difficulties
Status: Recruiting | Type: Observational
Sponsor: Masaryk University (Other)
Responsible Party: Sponsor
Other Study IDs: MUID2181034
Record Dates: First submitted 2025-06-11; First posted 2025-06-19 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Development Coordination Disorder; Motor Disabilities
Keywords: motor control; predictive control; feedback control; developmental coordination disorder -DCD; anticipatory postural adjustments- APA; interception task; preschool children; MABC-2; center of pressure - COP
MeSH Terms: conditions — Motor Skills Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- 1. Typical Development, Age 4.5-5.0: Preschool boys aged 4.5 to 5.0 years with typical motor development, as determined by scoring between the 16th and 84th percentile on the Movement Assessment Battery for Children - Second Edition (MABC-2). Participants will perform a catching task under two timing conditions while standing on a pressure mat and being video-recorded for motion analysis.
- 2. Typical Development, Age 6.5-7.0: Preschool boys aged 6.6 to 7.0 years with typical motor development, identified by MABC-2 scores between the 16th and 84th percentile. Children will complete the same experimental task involving the interception of a moving pendulum, with analysis of anticipatory postural adjustments and kinematics.
- 3. At Risk of DCD, Age 4.5-5.0: Preschool boys aged 4.5 to 5.0 years identified as at risk for Developmental Coordination Disorder (DCD), based on MABC-2 scores below the 16th percentile. Participants will perform a motor task catching a horizontally moving object under two time-constrained conditions, with simultaneous pressure and video data collection.
- 4. At Risk of DCD, Age 6.5-7.0: Preschool boys aged 6.6 to 7.0 years identified as at risk for motor coordination difficulties (DCD), based on scoring below the 16th percentile on the MABC-2. The experimental procedure includes a pendulum-catching task with detailed analysis of motor control and postural strategies.

SUMMARY:
This research project investigates the development of predictive and online motor control in preschool-aged boys with typical development and those with motor difficulties, specifically children at risk for Developmental Coordination Disorder (DCD). The study is being conducted as part of a doctoral dissertation at the Faculty of Sports Studies, Masaryk University in Brno, in cooperation with the integration and rehabilitation center Lentilka in Pardubice.

The aim of the study is to assess how children plan, initiate, and adjust their movements in response to a dynamic, time-sensitive task-catching a horizontally moving object (pendulum) under two different time constraints. By comparing performance between typically developing children and those identified as being at risk for motor difficulties, the study aims to improve our understanding of motor control development and support the creation of more effective diagnostic and educational strategies.

Participants in this study will be preschool boys from two age groups: 4.6 to 5.0 years and 6.5 to 7.0 years. Each age group will include 10 children with typical motor development and 10 children with motor difficulties, defined as scoring below the 16th percentile on the Movement Assessment Battery for Children - Second Edition (MABC-2). In total, the study aims to recruit 40 participants. Children with intellectual disabilities, autism spectrum disorder, uncorrected visual impairments, hearing loss, psychiatric or neurological conditions, or significant behavioral or orthopedic problems will be excluded from participation.

Each child will complete two parts of the study protocol. The first involves a standardized motor assessment using the MABC-2, which evaluates both fine and gross motor skills, including tasks such as threading beads, catching, and balance activities. The second part is an experimental task requiring interception of a swinging foam ring attached to a horizontal pendulum. The children will attempt to stop the pendulum at a precise moment under two time conditions: either on its first pass through the target zone (approximately 0.750 seconds after release) or on its second pass (approximately 1.5 seconds after release). The task will be performed using both the dominant and non-dominant hand, with multiple repetitions in each condition.

During the experiment, children will stand on a pressure-sensitive mat (CONFORMat® Tekscan), which records shifts in their center of pressure (COP). Upper limb movement will be captured using reflective markers placed on anatomical landmarks (shoulder, elbow, wrist, and hand), and recorded by four video cameras (two sagittal, two frontal). Movement data will be analyzed using Dartfish software.

The study will focus on several key outcome measures: anticipatory postural adjustments (APAs) based on COP movement prior to arm motion, spatial accuracy of the stopping movement (angular deviation), trajectory and velocity of COP displacement, timing of movement initiation based on radial styloid marker velocity, joint angles and segmental velocity, and overall smoothness of upper limb motion. All data and recordings will be pseudonymized, securely stored, and used exclusively for research purposes. Recordings will be deleted upon project completion.

This study aims to clarify the developmental trajectory of anticipatory and online motor control strategies in early childhood and to distinguish between typical and atypical motor patterns. The findings are expected to contribute to early screening practices and the development of targeted educational and therapeutic interventions for children with motor coordination difficulties. Ethical approval for the study has been granted by the Research Ethics Committee of Masaryk University. Participation is voluntary, and parents will receive individualized feedback on their child's motor performance after assessment.

DETAILED DESCRIPTION:
This study investigates the development of predictive and feedback motor control mechanisms in preschool-aged children (ages 4.5 to 7) during a visuomotor interception task. The primary objective is to evaluate age-related changes in upper limb coordination and postural control by comparing typically developing children with peers exhibiting motor difficulties, specifically those at risk for Developmental Coordination Disorder (DCD).

Interceptive actions, such as catching a moving object, impose high demands on the motor control system, requiring rapid integration of sensory information-visual and proprioceptive-alongside anticipatory postural adjustments and online movement corrections. In typically developing children, the capacity to anticipate and adapt to dynamic stimuli improves significantly between the ages of 4.5 and 7. In contrast, children with DCD often display impairments in these areas, which may be associated with deficits in internal modeling, reduced anticipatory postural adjustments (APAs), and delayed sensorimotor integration. To explore these mechanisms in a controlled environment, the study employs a dynamic bimanual interception task that involves stopping a foam circular pendulum moving horizontally along a rod. This setup allows for precise evaluation of motor response timing and quality, encompassing both upper limb kinematics and center of pressure (COP) displacement.

The research is based on a cross-sectional experimental design involving 60 preschool boys aged 4 to 7 years. Participants are evenly divided into three age cohorts and two motor proficiency groups, identified via the standardized Movement Assessment Battery for Children - Second Edition (MABC-2). Children scoring below the 16th percentile are classified as having motor difficulties. During the experiment, each child performs a bimanual interception task requiring them to stop the pendulum at a defined spatial target ("zero point") under two temporal conditions: intercepting the pendulum on its first pass (short interval, approximately 750 milliseconds from release) and on its second pass (long interval, approximately 1500 milliseconds from release). Multiple trials are conducted in each condition.

Upper limb movements are recorded using four high-resolution video cameras (sampling rate 50 Hz) positioned in sagittal and frontal planes. Motion is tracked via reflective markers placed on anatomical landmarks: the radial styloid process (wrist), lateral epicondyle (elbow), and deltoid insertion (shoulder). Postural control is assessed using a CONFORMat® pressure-sensitive platform operating at 100 Hz, which captures center of pressure trajectory and parameters relevant to anticipatory postural activity, including displacement, velocity, and root mean square (RMS) values. System synchronization is ensured through LED light pulses and color-coded timestamps, with an estimated precision of ±8 milliseconds. Video recordings are analyzed using Dartfish software, which is validated for 2D motion analysis, showing strong reliability (validity r ≥ .95; ICC ≥ .91).

Kinematic parameters include the timing of movement initiation relative to pendulum motion, peak velocity and time to peak velocity of the wrist marker, smoothness of the trajectory derived from acceleration profiles, and spatial accuracy of interception measured as angular deviation from the target. Postural variables include total COP path length as an indicator of stability, the range of movement in the anteroposterior and mediolateral directions, and the mean and RMS values of velocity and displacement during anticipatory postural phases.

This integrative approach allows for a detailed analysis of how young children plan, execute, and adapt their movements in real time. By comparing typically developing children with those at risk for motor coordination difficulties, the study aims to contribute to a better understanding of early motor control mechanisms and inform the development of more targeted diagnostic and intervention strategies.

ELIGIBILITY:
Inclusion Criteria:

* Age between 4.0 and 7.0 years (preschool age)
* Male sex
* Motor performance within the defined inclusion range based on the Movement Assessment Battery for Children - 2nd Edition (MABC-2)
* Typically developing children (as assessed by educators or therapists), or
* Children identified as having motor coordination difficulties

Exclusion Criteria:

* Children with intellectual disability
* autism spectrum disorder
* uncorrected vision impairment
* hearing loss
* neurological or psychiatric conditions, behavioral disorders, or orthopedic limitations will be excluded.

Ages: 4 Years to 7 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes
Study Population: The study population consists of preschool boys aged 4.5 to 7.0 years. Participants will be recruited from mainstream kindergartens and from an integrative preschool and rehabilitation center in the Czech Republic. The sample includes children with typical motor development, as well as children identified by educators and therapists as having motor coordination difficulties. Data will be collected within familiar educational or therapeutic environments to support natural task engagement.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-03-31 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Mean Onset Time of Upper-Limb Movement and Anticipatory Postural Adjustments (via COP) in a Horizontal Catching Task | single 60-minute session

CONTACTS AND LOCATIONS:
Locations (1):
- Lentilka - integrated kindergarden and rehabilitation center, Pardubice, Česká Republika, Czechia

REFERENCES:
- [Background] Gaveau V, Pisella L, Priot AE, Fukui T, Rossetti Y, Pelisson D, Prablanc C. Automatic online control of motor adjustments in reaching and grasping. Neuropsychologia. 2014 Mar;55:25-40. doi: 10.1016/j.neuropsychologia.2013.12.005. Epub 2013 Dec 13. PMID 24334110